CLINICAL TRIAL: NCT06923956
Title: Single Dose Oral Bioequivalence Study of Bempedoic Acid 180 mg Film Coated Tablet and Nilemdo® (Bempedoic Acid) 180 mg Film-coated Tablets in Healthy Adult Human Subjects Under Fasting Conditions.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C1B04874
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Hypercholesterolaemia; Mixed Dyslipidaemia; Cardiovascular Diseases
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bempedoic Acid Film Coated Tablet (Experimental): Bempedoic Acid 180 mg Film Coated Tablet
  Interventions: Drug: Bempedoic Acid Film Coated Tablet
- Nilemdo® (Bempedoic Acid) Film-coated tablets (Active Comparator): Nilemdo® (Bempedoic Acid) 180 mg Film-coated tablets
  Interventions: Drug: Nilemdo® (Bempedoic Acid) Film-coated tablets

INTERVENTIONS:
Drug: Bempedoic Acid Film Coated Tablet — 1 tablet of 180 mg Bempedoic Acid
  Arms: Bempedoic Acid Film Coated Tablet
Drug: Nilemdo® (Bempedoic Acid) Film-coated tablets — 1 tablet of 180 mg Bempedoic Acid
  Arms: Nilemdo® (Bempedoic Acid) Film-coated tablets

SUMMARY:
Single dose oral bioequivalence study of Bempedoic Acid 180 mg Film Coated Tablet and Nilemdo® (Bempedoic Acid) 180 mg Film-coated tablets in healthy adult human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 55 years old, both inclusive.
* Gender: Male and/or non-pregnant, non-lactating female.
* Female of child-bearing potential must have a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test performed within 28 days prior to first dosing day. They must be using an acceptable form of contraception.

For female of child-bearing potential, acceptable forms of contraception include the following:

* Non hormonal intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or
* Barrier methods containing or used in conjunction with a spermicidal agent, or
* Surgical sterilization or
* Practicing sexual abstinence throughout the course of the study.
* Female will not be considered of child-bearing potential if one of the following is reported and documented on the medical history:
* Postmenopausal with spontaneous amenorrhea for at least one year, or
* Spontaneous amenorrhea for more than 6 months and less than one year with Serum Follicular Stimulating Hormone (FSH) level > 40 mIU/mL, or
* Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or
* Total hysterectomy and an absence of bleeding for at least 3 months.
* BMI: 18.5 to 30.0 kg/m2, both inclusive; BMI value should be rounded off to one significant digit after decimal point (e.g. 30.04 rounds down to 30.0, while 18.45 rounds up to 18.5).
* Non-smokers and non-tobacco user (i.e. having no past history of smoking and tobacco consuming for at least one year prior to study).
* Able to communicate effectively with study personnel.
* Willing to provide written informed consent to participate in the study.
* All volunteers must be judged by the principal or sub-investigator or physician as normal and healthy during a pre-study safety assessment performed within 28 days of the first dose of study medication which will include:

Exclusion Criteria:

* History of allergic responses to Bempedoic acid or other related drugs, or any of its formulation ingredients.
* Have significant diseases or clinically significant abnormal findings during screening [medical history, physical examination (clinical examination), laboratory evaluations, ECG recording, gynecological history and examination (including pelvic examination and routine breast examination) (for female volunteers)].
* Any disease or condition like diabetes, psychosis or others, which might compromise the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system or any other body system.
* History or presence of bronchial asthma.
* Use of any hormone replacement therapy within 3 months prior to the first dose of study medication.
* Use of any depot injection or implant of any drug within 3 months prior to the first dose of study medication.
* Use of CYP enzyme inhibitors or inducers within 30 days prior to the first dose of study medication (see https://drug-interactions.medicine.iu.edu/MainTable.aspx).
* History or evidence of drug dependence or of alcoholism or of moderate alcohol use.
* History of difficulty with donating blood or difficulty in accessibility of veins.
* A positive hepatitis screen (includes subtypes B & C).
* A positive test result for HIV antibody.
* Volunteer who have received a known investigational drug within seven elimination half-life of the administered drug prior to the first dose of study medication.
* Volunteer who have donated blood or loss of blood 50 ml to 100 ml within 30 days or 101 ml to 200 ml within 60 days or >200 ml within 90 days (excluding volume drawn at screening for this study) prior to first dose of study medication, whichever is greater.
* History of difficulty in swallowing or of any gastrointestinal disease, which could affect drug absorption.
* Intolerance to venipuncture
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the principal investigator or sub-investigator, could contraindicate the volunteer's participation in this study.
* Institutionalized volunteer.
* Use of any prescribed medications (including simvastatin and pravastatin) within 14 days prior to the first dose of study medication.
* Use of any OTC products, vitamin and herbal products, etc., within 7 days prior to the first dose of study medication.
* Use of grapefruit and grapefruit containing products within 7 days prior to the first dose of study medication.
* Ingestion of any caffeine or xanthine products (i.e. coffee, tea, chocolate, and caffeinecontaining sodas, colas, etc.), recreational drugs, alcohol or other alcohol containing products within 48 hours prior to the first dose of study medication.
* Ingestion of any unusual diet, for whatever reason (e.g.: low sodium) for three weeks prior to the first dose of study medication.
* Volunteer having serum uric acid higher than the upper limit of normal range during screening.
* AST, ALT values are 1.1 times higher than the upper limit of normal range during screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Maximum measured plasma concentration over the time span specified (Cmax) | 72.00 hours
  The 90% confidence interval of the relative mean (geometric least square mean) of the test to reference product for Ln-transformed Pharmacokinetic parameters Cmax was to be within 80.00% to 125.00% for Bempedoic Acid to establish bioequivalence.
The area under the plasma concentration versus time curve was calculated using the linear trapezoidal linear interpolation rule from the zero time point to the last quantifiable concentration (AUCt) | 72.00 hours
  The 90% confidence interval of the relative mean (geometric least square mean) of the test to reference product for Ln-transformed Pharmacokinetic parameters AUCt was to be within 80.00% to 125.00% for Bempedoic Acid to establish bioequivalence.

SECONDARY OUTCOMES:
The area under the plasma concentration versus time curve from zero to infinity was calculated by adding Ct/Kel to AUCt, where Ct was the last quantifiable concentration and Kel was the elimination rate constant (AUCi) | 72.00 hours
  Descriptive statistics
Time of the maximum measured plasma concentration. If the maximum plasma concentration occurs at more than one time point, the first was chosen as Tmax (Tmax) | 72.00 hours
  Descriptive statistics
The terminal elimination rate constant was obtained from the slope of the line, fitted by linear least squares regression, through the terminal points of the natural log of the concentration versus time plot for these points (Kel) | 72.00 hours
  Descriptive statistics
The half-life was calculated by the equation tHalf = 0.693/ Kel (tHalf) | 72.00 hours
  Descriptive statistics

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research Limited, Noida, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No